CLINICAL TRIAL: NCT04420507
Title: Different Characteristics of Gut and Oral Microbiota of Women With Gestational Diabetes Mellitus
Brief Title: Gut and Oral Microbiome of GDM Patients During Pregnancy
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: Gut and oral microbiome of GDM
Record Dates: First submitted 2018-09-10; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-03

CONDITIONS: Gestational Diabetes; Pregnancy Related
Keywords: Gastrointestinal Microbiome; pregnancy; gestational diabetes mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stool samples were collected from objects in 3 time points：the first trimester(9-14 gestational weeks), the second trimester(24-28 gestational weeks) and the third trimester(32-37 gestational weeks). All the samples were collected at home by the participants using a PSP Spin Stool DNA kit, and the genomic DNA was extracted. The researchers only amplified the hypervariable V4 region of the bacterial 16S rRNA genes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GDM group: pregnant women who are diagnosed after 75g OGTT test between 24~27+6 gestational weeks
- health group: pregnant women who pass the 75g OGTT test and aren't diagnosed as GDM, and also don't have any other conditions, like hypertensive disorders, IBD, gastrointestinal ulcer, and so on.

SUMMARY:
The study aimed to clarify the characteristics of the intestinal and oral microbiome of Gestational Diabetes Mellitus(GDM) patients during the whole pregnancy, try to clarify the relationship between the microbiome and GDM.

DETAILED DESCRIPTION:
The aims of the study are to reveal the possibly natural change of the gut and oral microbiome of GDM patients during pregnancy, and to explorer whether GDM happened during pregnancy are associated with the maternal gut and oral microbiomes. As a perspective cohort study, the researchers will recruit pregnant women in early pregnancy（before 13 gestational weeks）and following the pregnancies till delivery. The stool samples and saliva samples of the recruits will be collected in 9~14,24~28 and 32~37 gestational weeks separately. The investigators will also perform oral examination between 24~28 weeks and sample subgingival plaque for test. Overall, all samples will be examined use 16S rRNA gene sequencing to analyze microbiome. And part of the samples of GDM patients will be analyzed using metagenomics. Combine with the pregnancy outcomes, the differences of gut and oral microbiome between GDM patients and healthy women will be expected, as well as the natural change during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* gestational age: before 13+6 weeks
* regular prenatal care in PUMCH

Exclusion Criteria:

* have medical history or current conditions： Gastrointestinal disorders, for example: Gastritis, gastric ulcer, inflammatory bowel disease; Hypertension; Diabetes; SLE or other severe CTD;
* pregnant, combine with malignancy diseases;
* pregnant, can't ensure regular prenatal check.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women who can ensure a regular prenatal check in the PUMCH OB clinic.
Sampling Method: Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
the gut and oral microbiome of GDM patients during pregnancy | the first trimester（9-14 gestational weeks), the second trimester (24-28 gestational weeks) and the third trimester(32-37 gestational weeks)
  The composition and species of gut and oral microbiome of GDM patients,separately in the first trimester（9-14 gestational weeks), the second trimester (24-28 gestational weeks) and the third trimester(32-37 gestational weeks).
the gut and oral microbiome of healthy pregnant women | the first trimester（9-14 gestational weeks), the second trimester (24-28 gestational weeks) and the third trimester(32-37 gestational weeks)
  The composition and species of gut and oral microbiome of healthy pregnant women ,separately in the first trimester（9-14 gestational weeks), the second trimester (24-28 gestational weeks) and the third trimester(32-37 gestational weeks).

SECONDARY OUTCOMES:
The glucose level during pregnancy | the first trimester（9-14 gestational weeks), the second trimester (24-28 gestational weeks) and the third trimester(32-37 gestational weeks)
  The fasting blood glucose level and the glycosylated albumin level in the first trimester（9-14 gestational weeks), the second trimester (24-28 gestational weeks) and the third trimester(32-37 gestational weeks). And the result of 75gOGTT test.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Edwards SM, Cunningham SA, Dunlop AL, Corwin EJ. The Maternal Gut Microbiome During Pregnancy. MCN Am J Matern Child Nurs. 2017 Nov/Dec;42(6):310-317. doi: 10.1097/NMC.0000000000000372. PMID 28787280
- [Result] Walker RW, Clemente JC, Peter I, Loos RJF. The prenatal gut microbiome: are we colonized with bacteria in utero? Pediatr Obes. 2017 Aug;12 Suppl 1(Suppl 1):3-17. doi: 10.1111/ijpo.12217. Epub 2017 Apr 26. PMID 28447406
- [Result] Jordan S, Baker B, Dunn A, Edwards S, Ferranti E, Mutic AD, Yang I, Rodriguez J. Maternal-Child Microbiome: Specimen Collection, Storage, and Implications for Research and Practice. Nurs Res. 2017 Mar/Apr;66(2):175-183. doi: 10.1097/NNR.0000000000000201. PMID 28252577
- [Result] Sharon G, Sampson TR, Geschwind DH, Mazmanian SK. The Central Nervous System and the Gut Microbiome. Cell. 2016 Nov 3;167(4):915-932. doi: 10.1016/j.cell.2016.10.027. PMID 27814521